CLINICAL TRIAL: NCT05889143
Title: A Prospective, Non-Intervention, Multi-Center Observational Study to Evaluate the Efficacy and Safety of CREZET Tablet in Patients With Dyslipidemia
Brief Title: A Study to Evaluate the Efficacy and Safety of CREZET Tablet
Status: Active, not recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWCRZ_OS_01
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mucotra® SR Tab
  Interventions: Drug: Ezetimibe/Rosuvastatin

INTERVENTIONS:
Drug: Ezetimibe/Rosuvastatin — Patient treated with Crezet Tablet
  Other Names: Crezet Tablet

SUMMARY:
This observation study is to evaluate blood lipid-lowering effects and liver/renal safety, changes in HbA1c and FPG in patients with dyslipidemia who administered CREZET tablets for 24 weeks.

DETAILED DESCRIPTION:
A subject who is diagnosed with dyslipidemia and scheduled to administer CREZET tablets, will be enrolled in this study based on the doctor's medical decision.

The CREZET Tablet will be administered for 24 weeks, and the data including demographic information, body measurement, vital signs and etc will be collected during the study period.

The data collection point is as follows.

1. Visit 1 (baseline, day 0)
2. Visit 2 (at 12 weeks)
3. Visit 3 (at 24 weeks)

ELIGIBILITY:
Inclusion Criteria:

1. an adult male and female over 19 years of age
2. A patient with dyslipidemia who is scheduled to administer Crezet tablets according to the medical judgment of the investigator based on permission
3. A person who voluntarily participates in the observational study and agrees in writing to comply with the subject's precautions during the study period after hearing and understanding the detailed explanation of the characteristics of the observational study and the drug to be studied

Exclusion Criteria:

1. A person who is prohibited from administering according to the permission of the Crezet definition

   * Patients who overreact to the principal or component of the Crezet definition
   * Patients with active liver disease or patients with persistent high symptoms of serum aminotransferase levels
   * a patient with a muscle disease
   * a patient administered in combination with a cyclosporine-med
   * Patients with severe renal failure (Creatinine Clearance (CLcr) < 30 mL/min)
   * Women and lactating women who may be pregnant or pregnant
   * Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
2. A person who has a history of taking Crezet tablets within three months of the date of registration
3. A person who is deemed inappropriate to participate in this observational study based on the judgment of investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of test subjects was calculated using the confidence interval of the rate of change, noting that the primary purpose of this observation study was to evaluate the rate of change in a single group.
  Recruitment of 14,151 people, which is 1.5%, was expected by referring to the minimum number of subjects required and the estimated patients taking two components of single drug and ezetimib compound.
  However, this study was a non-intervention observation study conducted under daily treatment, and it was confirmed that the number of subjects who applied 10% of the dropout rate was about 15,000 Therefore, this study will be conducted with study population of 15,000 subjects.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The Rate of change in LDL-C | 24 weeks
  The Rate of change in LDL-C at 24 weeks from baseline

SECONDARY OUTCOMES:
The Rate of change in LDL-C | 12 weeks
  The Rate of change in LDL-C at 12 weeks from baseline
The change in HbA1c | 12 weeks
  The change in HbA1c at 12 weeks from baseline
The change in HbA1c | 24 weeks
  The change in HbA1c at 24 weeks from baseline
The change in FPG | 12 weeks
  The change in FPG at 12 weeks from baseline
The change in FPG | 24 weeks
  The change in FPG at 24 weeks from baseline
The chanage in lipid variable | 12 weeks
  The chanage in lipid variable at 12 weeks from baseline
The chanage in lipid variable | 24 weeks
  The chanage in lipid variable at 24 weeks from baseline
The change in AST | 12 weeks
  The change in AST at 12 weeks from baseline
The change in AST | 24 weeks
  The change in AST at 24 weeks from baseline
The change in ALT | 12 weeks
  The change in ALT at 12 weeks from baseline
The change in ALT | 24 weeks
  The change in ALT at 24 weeks from baseline
Percentage of subjects who reached LDL-C target | 12 weeks
  Percentage of subjects who reached LDL-C target according to Korean Society of Lipid Arteriosclerosis's risk classification of treatment guidelines for dyslipidemia at 12 weeks from baseline
Percentage of subjects who reached LDL-C target | 24 weeks
  Percentage of subjects who reached LDL-C target according to Korean Society of Lipid Arteriosclerosis's risk classification of treatment guidelines for dyslipidemia at 24 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: JunYoung Park, Study Director — Daewoong Pharma
Locations (1):
- Kimyounggi Clinic, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this point